CLINICAL TRIAL: NCT02795364
Title: A Prospective Study About the Validity of MRS-guided Resection on Prognosis High-grade Gliomas
Brief Title: Study About the Validity of MRS-guided Resection on Prognosis High-grade Glioma Gliomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2016-232
Record Dates: First submitted 2016-05-24; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Glioma; Anaplastic Oligoastrocytoma; Glioblastomas (GBM)
Keywords: High Grade Glioma; Magnetic Resonance Spectroscopy; Surgical resection; Prognosis
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structural Image Guidance (Active Comparator): In this arm, the patients will receive maximum resection of the tumor with the MRI T1W-enhanced image guidance, in addition to the standard therapy
  Interventions: Procedure: Structural Image Guidance
- Metabolic Image Guidance (Experimental): In this arm, the patients will receive quantitative resection of the tumor with both the MRI T1W-enhanced and the MRS Cho-to-NAA index (CNI) image guidance, in addition to the standard therapy.
  Interventions: Procedure: Metabolic Image Guidance

INTERVENTIONS:
Procedure: Structural Image Guidance — Resecting the tumor in accordance with the margin on MRI T1W-enhanced delineation
  Arms: Structural Image Guidance
Procedure: Metabolic Image Guidance — Aggressive resecting of the tumor in accordance with the margin on MRS CNI delineation
  Arms: Metabolic Image Guidance

SUMMARY:
Gliomas,especially high-grade glioma ,are the most common primary malignant brain tumor in adults,yet outcomes from this aggressive neoplasm remain dismal.The extent of resection is one of the most essential factors that influence the outcomes of glioma resection.However, conventional structural imaging has failed to accurately delineate glioma margins because of tumor cell infiltration. the investigators have finished few project that suggest the feasibility of Magnetic Resonance Spectrum(MRS)-guided resection,unfortunately, lacking sufficient clinical evidence.This prospective cohort study is to provide a clinical evidence for the validity of MRS-guided resection in patients with HGG .

DETAILED DESCRIPTION:
High-grade glioma(HGG), including anaplastic glioma (AG) and Glioblastomas (GBM), are associated with poor prognosis, even with all the scientific development of the last decades, attributed to optimally treated with maximum safe surgery, followed by radiotherapy (RT) and/or systemic chemotherapy (CT). Despite recent advances in treatment, the prognosis of HGG remains poor with comparatively short overall survival (OS) and importantly profound impact on quality of life (QoL).Admittedly,multiple factors are related to their outcome, including age, biological characteristics of the tumor, and extent of treatment. Notably, extent of resection (EOR) plays a major role as an independent modifiable factor associated with improved overall and progression-free survival. Achievement of maximal safe resection, removing as much as possible the tumor while preserving the neurological function, is the main goal of the current surgical treatment of High-grade glioma (HGG).

Many researchers took into study about the extent of surgery ,despite exist various editions,produced similar results, although only one randomized controlled trial(RCT) provided 1-year PFS data and there was no significant difference between total resection and incomplete resection in that study. It suggests that should push the delineation of tumour outward for better prognosis.therefore,the core of conservation point to the simon-pure margins that proximate to histopathologic periphery of HGG.Consequently, analyses showed that the resection of ≥ 53.21% of the surrounding FLAIR abnormality beyond the 100% contrast-enhancing resection was associated with a significant prolongation of survival compared with that following less extensive resections,neo-FLAIR abnormality region is gradually coming into people' vision,supportive evidence is warranted for the relationship of extensive resection and reasonable prognosis,which equal to draw the scope of tumour margins that has been put forward to sketch via metabolic information.

During previous clinical practice,the investigators have researched that the correlation of metabolic information and tumour identification about true-false type,study suggests that Cho/tNAA ratio threshold values of 0.5, 1.0, 1.5 and 2.0 appeared to predict the specie-mens containing the tumour with respective probabilities of 0.38, 0.60, 0.79, 0.90 in HGG and 0.16, 0.39, 0.67, 0.87 in LGG,it is interesting to reveal the metabolic action of true-tumour,and immediately the other work projected by our group found that the differences between the structural and the metabolic volumes with Cho/tNAA ratio(CNI) thresholds of 0.5 and 1.5 were statistically significant (p = 0.0005 and 0.0129, respectively) and 0.5 and 1.0 were statistically significant in HGG.Problem,whether operation that resect by delineation at Cho/tNAA ratio threshold 1.0 can bring better outcome ,remains to be solved,namely,the investigators need further clinical evidence .

Based on this thoughtfulness, this prospective cohort study is to provide a reasonable evidence for the correlation between metabolic-guide resection and the prognosis of the HGGs , cohorts contain 25 cases in the arm group and 25 cases in the control group.Respectively receive different operation project followed by statistical analysis aim at overall survival (OS)and progression free survival (PFS).Definitively,the investigators hope to draw a conclusion that armed group has better outcome,like that,studies have a step in the course of HGG therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age ≤ 70 years, both genders.
* Post-operative histological pathology confirms HGGs (anaplastic glioma (AG) and Glioblastomas (GBM),2007 World Health Organization(WHO) classification Grade III IV).
* No chemotherapy and radiotherapy history
* Karnofsky performance score of ≥ 60%
* Written informed consent must be obtained from all patients, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Tumor involves more than 3 cerebral lobes (gliomatosis or multiple gliomas ).
* Tumor is histopathology verified or complicated with other intracranial neoplasms (e.g. metastatic tumors ).
* Tumor is complicated with systematic malignancies.
* Tumor recurrence or complicated with disease that result in psychological and cognitive problem
* Participate in other clinical trials at meantime.
* Voluntarily quit .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | within 1 year after the surgery
  To determine time to death in the enrolled patients.

SECONDARY OUTCOMES:
Progression free survival (PFS) | within 1 year after the surgery
  The survival rate of followed patients without progressive disease (PD) 3, 6, 9, and 12 months after the operation,To determine time to tumor progression in this The survival rate of followed patients without progressive disease (PD) 3,6, 9,and 12 months after the operation,To determine time to tumor progression in this patient population
Karnofsky performance status (KPS) | 3, 6, 9 and 12 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, Professor, Principal Investigator — Huashan Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Le Rhun E, Rhun EL, Taillibert S, Chamberlain MC. The future of high-grade glioma: Where we are and where are we going. Surg Neurol Int. 2015 Feb 13;6(Suppl 1):S9-S44. doi: 10.4103/2152-7806.151331. eCollection 2015. PMID 25722939
- [Background] Mohammadi AM, Hawasli AH, Rodriguez A, Schroeder JL, Laxton AW, Elson P, Tatter SB, Barnett GH, Leuthardt EC. The role of laser interstitial thermal therapy in enhancing progression-free survival of difficult-to-access high-grade gliomas: a multicenter study. Cancer Med. 2014 Aug;3(4):971-9. doi: 10.1002/cam4.266. Epub 2014 May 9. PMID 24810945
- [Background] Li XZ, Li YB, Cao Y, Li PL, Liang B, Sun JD, Feng ES. Prognostic implications of resection extent for patients with glioblastoma multiforme: a meta-analysis. J Neurosurg Sci. 2017 Dec;61(6):631-639. doi: 10.23736/S0390-5616.16.03619-5. Epub 2016 Jan 29. PMID 26824196
- [Background] Li YM, Suki D, Hess K, Sawaya R. The influence of maximum safe resection of glioblastoma on survival in 1229 patients: Can we do better than gross-total resection? J Neurosurg. 2016 Apr;124(4):977-88. doi: 10.3171/2015.5.JNS142087. Epub 2015 Oct 23. PMID 26495941
- [Background] Guo J, Yao C, Chen H, Zhuang D, Tang W, Ren G, Wang Y, Wu J, Huang F, Zhou L. The relationship between Cho/NAA and glioma metabolism: implementation for margin delineation of cerebral gliomas. Acta Neurochir (Wien). 2012 Aug;154(8):1361-70; discussion 1370. doi: 10.1007/s00701-012-1418-x. Epub 2012 Jun 23. PMID 22729482
- [Background] Zhang J, Zhuang DX, Yao CJ, Lin CP, Wang TL, Qin ZY, Wu JS. Metabolic approach for tumor delineation in glioma surgery: 3D MR spectroscopy image-guided resection. J Neurosurg. 2016 Jun;124(6):1585-93. doi: 10.3171/2015.6.JNS142651. Epub 2015 Dec 4. PMID 26636387
- [Background] Zou QG, Xu HB, Liu F, Guo W, Kong XC, Wu Y. In the assessment of supratentorial glioma grade: the combined role of multivoxel proton MR spectroscopy and diffusion tensor imaging. Clin Radiol. 2011 Oct;66(10):953-60. doi: 10.1016/j.crad.2011.05.001. Epub 2011 Jun 12. PMID 21663899
- [Background] Aibaidula A, Lu JF, Wu JS, Zou HJ, Chen H, Wang YQ, Qin ZY, Yao Y, Gong Y, Che XM, Zhong P, Li SQ, Bao WM, Mao Y, Zhou LF. Establishment and maintenance of a standardized glioma tissue bank: Huashan experience. Cell Tissue Bank. 2015 Jun;16(2):271-81. doi: 10.1007/s10561-014-9459-4. Epub 2014 Jun 15. PMID 24929994